CLINICAL TRIAL: NCT03219892
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Freezing of Gait in Parkinson's Disease
Brief Title: rTMS for the Treatment of Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Piu Chan, Director, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z171100000117013
Record Dates: First submitted 2017-07-03; First posted 2017-07-18 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Parkinson's Disease
Keywords: freezing of gait; rTMS; fMRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-frequency rTMS (Experimental): Patients randomized to this group will receive rTMS delivering over the supplementary motor area (SMA). Each treatment consists 1000 pulses (5-second burst of 10Hz rTMS, repeated 20 times at every minute ).Stimulus intensity is 90% of resting motor threshold. A figure-of-8 coil is connected to a biphasic magnetic stimulator, and the induced current is perpendicular to the midline.
  Interventions: Device: High-frequency rTMS
- Sham rTMS (Sham Comparator): Patients randomized to this group will receive the sham rTMS. The procedure is same as used in patients receiving experimental rTMS, except that the coil is angled 90° away.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: High-frequency rTMS — It is delivered at a 5-second burst of 10Hz stimuli, repeated 20 times at every minute. Each treatment contains a total of 1000 pulses. Stimulus intensity is 90% of resting motor threshold. The SMA stimulation will be given using a coil centered at points 3-cm anterior to the leg motor area in the sagittal midline.
  Arms: High-frequency rTMS
Device: Sham rTMS — The procedure will be same as the high-frequency rTMS except that the coil is 90° angled away.
  Arms: Sham rTMS

SUMMARY:
This study is a double blind comparative study examining the effectiveness of the rTMS treatment on Freezing of Gait (FOG) in patients with Parkinson's disease (PD). The investigators hypothesize that treatment with rTMS on supplemental motor area will improve gait quality and decrease the frequency of FOG in PD patients.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is a common and debilitating symptom in patients with Parkinson's disease (PD), characterized by sudden and brief episodes of inability to produce effective forward stepping. FOG is a major risk factor for falls, and greatly contributes to reduced mobility and quality of daily life. Treatment of FOG has been perceived as a very challenging task. Although various treatment approaches exist, including pharmacological and surgical options, evidence is inconclusive for many approaches and no clear treatment protocols are available until now.

Repetitive transcranial magnetic stimulation (rTMS), a noninvasive neural modulation technique, has been closely applied as a treatment for various neurologic and psychiatric disorders. A recent meta-analysis demonstrated that rTMS could improve motor symptoms for PD patients with a moderate effect size. To date, however, only few rTMS studies have focused on its efficacy on FOG in patients with parkinsonism, and most of them targeted the primary motor cortex or dorsolateral prefrontal cortex . Even though some evidence indicates the involvement of the SMA in FOG, no report has described the SMA rTMS in PD patients with FOG.

Moreover, few studies combined functional magnetic resonance imaging (fMRI) and rTMS to unravel the mechanism of its beneficial effects. To address these issues, the investigators conducted a randomized, double-blind, sham-controlled study to explore the efficiency of SMA-rTMS on FOG in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD patients.
* Presenting with FOG.
* The mini-mental state examination questionnaire score above 24 points.

Exclusion Criteria:

* Other neurological or psychiatric disorders.
* History of epilepsy, seizures or convulsions.
* Metal implantation.
* History of exposure to rTMS in the past (to minimizing risk of unblinding sham condition).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piu Chan, MD, PhD, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-frequency rTMS | Sham rTMS
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-frequency rTMS | Sham rTMS | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 24
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.65 (10.56) | 65.60 (8.68) | 63.63 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 9 | 5 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 20 | 10 | 30
Region of Enrollment [Number; unit: participants]
  China | 20 | 10 | 30
New Freezing of Gait Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Ranging from 0-24, with a higher score indicating a worse outcome.
  units on a scale | 15.85 (4.87) | 14.70 (4.03) | 15.34 (4.43)

OUTCOME MEASURES:

1. Primary Outcome: Changes of the New Freezing of Gait Questionnaire (NFOGQ) Score
Description: NFOGQ ranges from 0-24 points. It is used to quantify changes of the FOG frequency and severity. Higher scores mean a worse outcome.
Time Frame: Pre-treatment, post-treatment 4 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High-frequency rTMS | Sham rTMS
Number analyzed (Participants) | 20 | 10
score on a scale | -1.60 [-2.37 to -0.83] | -2.13 [-2.97 to -1.29]

2. Secondary Outcome: Motor Subscale of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS Part III)
Description: The motor subscale of the Movement Disorder Society Unified Parkinson's Disease Rating Scale evaluates the overall motor symptoms in PD, ranging from 0-112 points. Higher scores mean a worse outcome.
Time Frame: Pre-treatment, post-treatment 4 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High-frequency rTMS | Sham rTMS
Number analyzed (Participants) | 20 | 10
score on a scale | -5.79 [-7.86 to -3.71] | -0.24 [-3.17 to 2.69]

3. Secondary Outcome: Cadence
Description: To assess the changes of straight walking function.
Time Frame: Pre-treatment, post-treatment 4 weeks
Measure: Mean (95% Confidence Interval); unit: steps/minute
Arm/Group | High-frequency rTMS | Sham rTMS
Number analyzed (Participants) | 20 | 10
steps/minute | 2.67 [-1.27 to 6.61] | -7.99 [-13.68 to -2.30]

4. Secondary Outcome: Turning Duration
Description: To assess the changes of turning function.
Time Frame: Pre-treatment, post-treatment 4 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | High-frequency rTMS | Sham rTMS
Number analyzed (Participants) | 20 | 10
seconds | -0.47 [-0.89 to -0.05] | 0.59 [-0.55 to 0.71]

5. Secondary Outcome: Changes of Brain Functional Connectivity.
Description: functional connectivity will be assessed using fMRI, which can help understand the neural mechanism of the rTMS treatment. Using the baseline scans, the imaging biomarkers for freezing of gait and Parkinson's disease were developed by contrasting the connectivity profiles of patients with freezing of gait to those without freezing of gait and normal controls, respectively. These two biomarkers were then interrogated to assess the rTMS effects on connectivity patterns.
Time Frame: Pre-treatment, post-treatment at 2 weeks
Measure: Mean (Standard Deviation); unit: correlation coefficients
Arm/Group | High-frequency rTMS | Sham rTMS
Number analyzed (Participants) | 20 | 10
correlation coefficients
  before treatment | 0.33 (0.12) | 0.33 (0.18)
  after treatment | 0.49 (0.19) | 0.50 (0.18)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | High-frequency rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 3/20 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-frequency rTMS (N=20) | Sham rTMS (N=10)
mild but tolerable headache (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03219892/Prot_SAP_000.pdf